CLINICAL TRIAL: NCT01471470
Title: A Phase II Study of Neoadjuvant Chemotherapy With Docetaxel, Capecitabine, Cisplatin, and Bevacizumab in Patients With Unresectable Advanced Gastric Cancer
Brief Title: Efficacy of Docetaxel, Capecitabine, Cisplatin, and Bevacizumab in Patients With Unresectable Advanced Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Principal Investigator, Yoon-Koo Kang, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC1003
Record Dates: First submitted 2011-07-18; First posted 2011-11-15 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Advanced Gastric Cancer
Keywords: Advanced gastric cancer; Neoadjuvant; Bevacizumab
MeSH Terms: interventions — Docetaxel; Capecitabine; Cisplatin; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- neoadjuvant (Experimental)
  Interventions: Drug: Docetaxel, Capecitabine, Cisplatin, Bevacizumab

INTERVENTIONS:
Drug: Docetaxel, Capecitabine, Cisplatin, Bevacizumab — Bevacizumab 7.5mg/kg IV (D1) Docetaxel 60 mg/m2 IV (D1) Cisplatin 60 mg/m2 IV (D1) Xeloda 1,875 mg/m2/day/bid PO (D1-D14)

SUMMARY:
The purpose of this study is to determine whether docetaxel, capecitabine, cisplatin, and bevacizumab are effective in the treatment of unresectable advanced gastric cancer.

DETAILED DESCRIPTION:
In our previous phase II study of neoadjuvant docetaxel, capecitabine and cisplatin chemotherapy, patients with unresectable gastric cancer because of invasion to adjacent organs or metastasis to para-aortic lymph nodes received benefit from neoadjuvant chemotherapy. Based on these results and reports that bevacizumab enhances response rate, we planned docetaxel, capecitabine, cisplatin, and bevacizumab as neoadjuvant chemotherapy for patients with local invasion or para-aortic node metastasis alone.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented adenocarcinoma of the stomach or gastroesophageal junction.
* Invasion to adjacent organ (T4) proven by endoscopic ultrasonography (EUS) or presence of paraaortic lymph node metastasis by CT and PET(short-axis diameter > 1 cm showing hot uptake in PET scan).
* Age 18-70 years old
* ECOG performance status 0-2
* Adequate hepatic function(serum bilirubin <1.5mg/dl, AST (SGOT) and ALT (SGPT) < 2.5 x UNL, alkaline phosphatase < 5 x UNL)
* Adequate renal function(serum creatinine <1.5mg/dl)
* Adequate bone marrow function (WBC ≥4000 cell/㎕ with ANC ≥1500 cell/㎕, platelet count ≥100,000 cell/㎕)
* HER2 negative (HER2 immunohistochemistry 0 or 1+, immunohistochemistry 2+ but FISH negative)
* Informed consent

Exclusion Criteria:

* Other histologic type than adenocarcinoma
* Metastasis in other sites than paraaortic lymph nodes, like in liver or peritoneum.
* Presence or history of other cancers
* History of prior chemotherapy, antiangiogenic agents, or radiation.
* Patients with definite ascites in abdomen CT scan
* Presence of not adequately controlled CNS metastasis
* Bowel obstruction
* Evidence of gastrointestinal bleeding
* Other serious illness or medical conditions including hypertension uncontrolled by medication.
* Pregnant or lactating women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-07 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
R0 resection rate | Up to 4 weeks after surgery
  R0 resection means complete resection of tumor.

SECONDARY OUTCOMES:
Overall survival | Up to 3 years
  Overall survival will be measured from the start of study treatment to documented death of any cause.
Progression-free survival | Up to 3 years
  Time to progression will be measured from the start of study treatment to documented tumor progression.
Adverse Event | Up to 28 days after end of treatment
  Treatment toxicities are evaluated according to the NCI common toxicity criteria version 3.0
Angiogenetic biomarkers | Baseline and 6 weeks after treatment
  cluster of differentiation 31, microvessel density, platelet derived growth factor, vascular endothelial growth factor-A, vascular endothelial growth factor receptor-1, vascular endothelial growth factor receptor-2, Neuropilin 1 and phosphatidylinositol glycan anchor biosynthesis, class F

CONTACTS AND LOCATIONS:
Overall Officials: Yoon-Koo Kang, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea